CLINICAL TRIAL: NCT02623959
Title: A Double Blind Randomized Controlled Trial of Indwelling Pleural Catheters Versus Indwelling Pleural Catheters Plus Doxycycline Pleurodesis for Treatment of Malignant Pleural Effusions
Brief Title: Indwelling Pleural Catheter With Either Doxycycline or Saline at Day 7 for Pleurodesis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-0142; NCI-2016-00658 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Advanced Cancers; Malignant Pleural Effusions
Keywords: Advanced Cancers; Malignant pleural effusions; MPE; Indwelling pleural catheter; IPC; Questionnaires; Surveys; Fentanyl patch; Fentanyl by vein; Sublimaze; Doxycycline; Vibramycin; Periostat; Doryx; :Phone calls
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Surveys and Questionnaires; Fentanyl; Sodium Chloride; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Indwelling Pleural Catheter (IPC) + Saline (Experimental): Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Saline in the catheter.
  After the IPC is removed, participant is called one time each month by study staff to check on their status.
  Interventions: Behavioral: Questionnaires; Drug: Fentanyl Patch; Drug: Fentanyl (IV); Other: Saline; Behavioral: Phone Calls
- Indwelling Pleural Catheter (IPC) + Doxycycline (Active Comparator): Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Doxycycline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Doxycycline in the catheter.
  After the IPC is removed, participant is called one time each month by study staff to check on their status
  Interventions: Behavioral: Questionnaires; Drug: Fentanyl Patch; Drug: Fentanyl (IV); Drug: Doxycycline; Behavioral: Phone Calls

INTERVENTIONS:
Behavioral: Questionnaires — Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline or Doxycycline.
  Other Names: Surveys
Drug: Fentanyl Patch — Participant given a Fentanyl patch, 12 mcg/hour, which should be worn at follow up visit 5 days after IPC placement.
Drug: Fentanyl (IV) — Fentanyl 50 mcg given by vein prior to catheter draining.
  Other Names: Sublimaze
Other: Saline — Catheter is drained then Saline placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Arms: Indwelling Pleural Catheter (IPC) + Saline
Drug: Doxycycline — Catheter is drained then Doxycycline 500 mg placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Other Names: Vibramycin; Periostat; Doryx
  Arms: Indwelling Pleural Catheter (IPC) + Doxycycline
Behavioral: Phone Calls — After the IPC is removed, participant is called one time each month by study staff to check on their status.

SUMMARY:
The goal of this clinical research study is to compare indwelling pleural catheters (IPC) in combination with saline (the current standard of care) versus IPC in combination with doxycycline as treatment for pleural effusions.

DETAILED DESCRIPTION:
IPC Placement and Placement Follow-Up:

Before the IPC is inserted, you will complete 2 questionnaires about your quality of life and any symptoms you may have. It should take no more than 15-20 minutes to complete. You will also have a chest x-ray and you will rate your pain on a scale of 1-10. These tests are all part of your standard of care and can be explained to you in more detail by your doctor. You will be required to sign a separate consent form in order to have the IPC placed. Your doctor will give you detailed instructions about the IPC placement procedure, including its risks.

After the IPC is placed, the doctor will give you a prescription for a fentanyl patch to help control pain. The study staff will tell you how and when to wear the fentanyl patch and about any side effects that are associated with fentanyl.

About 5 days (+/- 2 days) after the IPC has been placed, you will have a clinic visit where you will be checked up on as part of your standard of care. It is important that you wear your fentanyl patch in the morning before this visit. At this clinic visit, the results of a previously performed chest x-ray will be reviewed, you will be asked to rate your pain on a scale of 1-10, and you will be asked how much fluid has drained from your catheter.

Based on the results of the above Day 5 check-up, if you are found to be ineligible to receive the study drug, the fentanyl patch will be taken off and you will be followed as part of your usual care. However, you will still considered to be on study and you will be followed the same as a participant who receives the study drug.

If you are found to be eligible to receive the study drug, you will receive fentanyl by vein over a few minutes, if needed to help control your pain. The study staff will then begin to drain your catheter and either doxycycline or saline (described below) will be placed in the catheter. The catheter will be capped for 1 hour and then drained again.

To determine if you will receive doxycycline or saline, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If you are in Group 1, you will receive doxycycline.
* If you are in Group 2, you will receive saline.

Neither you nor the study doctor will know if you are receiving doxycycline or saline. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Length of Study Participation:

You will receive doxycycline or saline 1 time on this study. Your participation on this study will be over if you withdraw consent or the study closes, whichever takes place first.

Follow-Up:

Between 10-14 days after you have received either doxycycline or saline, you will come to the clinic as part of your usual standard of care so the doctor can check your IPC for possible leaking, infection, to see how much fluid has drained, and to remove any sutures. The catheter may be removed if you have it is leaking or shows signs of infection. You will continue to have this visit 1 time each month as part of your standard of care until the catheter is removed. During each of these visits:

* You will have a chest x-ray to check the status of your lungs.
* You will complete the same 2 questionnaires that you completed before your IPC was placed.

Long-Term Follow-Up:

One (1) time each month after the IPC is removed, you will be called and asked how you are doing, if you are having any side effects, if the disease has come back, and about your overall quality of life. Some of this information may be collected from your medical record. Each phone call should last about 5-10 minutes.

This is an investigational study. Doxycycline is FDA approved and commercially available for the treatment of different types of infections and pleural effusions. It is considered investigational to compare doxycycline to saline to treat pleural effusions.

Up to 250 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with MPE undergoing IPC placement
2. Age 18 or older
3. Sufficient mental capacity to answer SF-6D and Borg score questions.

Exclusion Criteria:

1. Patients undergoing pleurodesis for benign disease (e.g., spontaneous pneumothorax)
2. Inability or unwillingness to give informed consent
3. Inability to perform phone call and clinical follow-up at MDACC
4. Previous intrapleural therapy for MPE on the same side
5. Chylous effusions associated with malignant disease
6. ECOG of 4 and life expectancy </= 2 weeks
7. Doxycycline allergy
8. Contraindication to placement of an IPC (e.g., uncorrected coagulopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ost, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients with MPE eligible for IPC,no evidence of extensive loculation or hydropneumothorax or other contraindication to pleurodesis or narcotics;aged 18 or older;and has sufficient mental capacity to answer SF-6D and Borg score questions. Out of 3 participants 2 withdrew before randomization.
Groups:
- Indwelling Pleural Catheters (Randomized to Saline): On Day 5, Fentanyl patch 12 mcg/hr placed if not already on, Fentanyl 50 mcg IV given, drain maximally, saline instilled, catheter capped for 1 hour and then re-drain. Pain will assess using a Visual Analogue Scale (VAS) as well, patient discharged home.
  Symptom and quality of life questionnaires will be completed at baseline, at 10 - 14 days and each month for 12 months as well as recurrence status defined as recurrent effusion on the same side requiring intervention will be documented.
- Indwelling Pleural Catheters+Doxycycline (Randomized to Rx Arm: On Day 5, Fentanyl patch 12 mcg/hr placed if not already on, Fentanyl 50 mcg IV given, drain maximally, doxycycline instilled, Catheter is capped for 1 hour and then re-drain. Pain will assess using a Visual Analogue Scale as well, patient discharged home.
  Symptom and quality of life questionnaires will be completed at baseline, at 10 - 14 days and each month for 12 months as well as recurrence status defined as recurrent effusion on the same side requiring intervention will be documented.
Period: Overall Study
Arm/Group | Indwelling Pleural Catheters (Randomized to Saline) | Indwelling Pleural Catheters+Doxycycline (Randomized to Rx Arm
Started | 0 | 1
Completed | 0 | 0 (due to progression)
Not Completed | 0 | 1
Not completed — Progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 participants withdrew before randomization
Groups:
- Indwelling Pleural Catheters (IPC) (Randomized to Saline): Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Saline in the catheter. After the IPC is removed, participant is called one time each month by study staff to check on their status. Questionnaires: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline or Doxycycline.
  Fentanyl Patch: Participant given a Fentanyl patch, 12 mcg/hour, which should be worn at follow up visit 5 days after IPC placement.
  Fentanyl (IV): Fentanyl 50 mcg given by vein prior to catheter draining.
  Saline: Catheter is drained then Saline placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Phone Calls: After the IPC is removed, partici
- IPC Plus Doxycycline (Randomized to Rx Arm): Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Doxycycline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Doxycycline in the catheter.
  After the IPC is removed, participant is called one time each month by study staff to check on their status. Questionnaires: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline or Doxycycline.
  Fentanyl Patch: Participant given a Fentanyl patch, 12 mcg/hour, which should be worn at follow up visit 5 days after IPC placement.
  Fentanyl (IV): Fentanyl 50 mcg given by vein prior to catheter draining.
  Doxycycline: Catheter is drained then Doxycycline 500 mg placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Phone Calls: After th
- Total: Total of all reporting groups
Arm/Group | Indwelling Pleural Catheters (IPC) (Randomized to Saline) | IPC Plus Doxycycline (Randomized to Rx Arm) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcomes of Interest Will be Time to Catheter Removal.
Description: This outcome will be analyzed by cause-specific hazard Cox model with treatment group as a covariate. Whenever a catheter is removed the cause for removal will be documented. For the analysis causes will include removal due to decreased drainage (i.e. as per plan) as well as removal due to complications (e.g. infection, empyema, and refractory pain) or other reasons (e.g. catheter plugged but no complication to the patient, patient preference without a complication).
Time Frame: 1 month
Population: Due to slow accrual and the design of the study the protocol was terminated. No data was collected and no analysis was done.
Groups:
- Indwelling Pleural Catheter (IPC) + Saline: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Saline in the catheter.
  After the IPC is removed, participant is called one time each month by study staff to check on their status.
  Questionnaires: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline or Doxycycline.
  Fentanyl Patch: Participant given a Fentanyl patch, 12 mcg/hour, which should be worn at follow up visit 5 days after IPC placement.
  Fentanyl (IV): Fentanyl 50 mcg given by vein prior to catheter draining. Saline: Catheter is drained then Saline placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Phone Calls: After the IPC is removed, partici
- Indwelling Pleural Catheter (IPC) + Doxycycline: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Doxycycline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Doxycycline in the catheter.
  After the IPC is removed, participant is called one time each month by study staff to check on their status Questionnaires: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline or Doxycycline.
  Fentanyl Patch: Participant given a Fentanyl patch, 12 mcg/hour, which should be worn at follow up visit 5 days after IPC placement.
  Fentanyl (IV): Fentanyl 50 mcg given by vein prior to catheter draining. Doxycycline: Catheter is drained then Doxycycline 500 mg placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Phone Calls: After th
Arm/Group | Indwelling Pleural Catheter (IPC) + Saline | Indwelling Pleural Catheter (IPC) + Doxycycline
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Assessment of Symptom Burden, Pleurodesis Efficacy, Complications, Health Care Resource Utilization, the Need of Hospitalization for Pain Control, Pain Free Days and Mortality
Time Frame: baseline and 1 month
Population: Due to slow accrual and the design of the study the protocol was terminated and no analysis was done.
Groups:
- Indwelling Pleural Catheters (Randomized to Saline): Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Saline in the catheter. After the IPC is removed, participant is called one time each month by study staff to check on their status. Questionnaires: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline or Doxycycline.
  Fentanyl Patch: Participant given a Fentanyl patch, 12 mcg/hour, which should be worn at follow up visit 5 days after IPC placement.
  Fentanyl (IV): Fentanyl 50 mcg given by vein prior to catheter draining.
  Saline: Catheter is drained then Saline placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Phone Calls: After the IPC is removed, partici
- Indwelling Pleural Catheters Plus Doxycycline (Randomized to R: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Doxycycline. Participant given a Fentanyl patch which should be worn at follow up visit 5 days after IPC placement. Fentanyl patch then be removed and Fentanyl by vein given prior to catheter draining. Study staff drains the IPC and places Doxycycline in the catheter.
  After the IPC is removed, participant is called one time each month by study staff to check on their status. Questionnaires: Symptom and quality of life questionnaires completed at baseline and at 10 - 14 days after receiving Saline or Doxycycline.
  Fentanyl Patch: Participant given a Fentanyl patch, 12 mcg/hour, which should be worn at follow up visit 5 days after IPC placement.
  Fentanyl (IV): Fentanyl 50 mcg given by vein prior to catheter draining.
  Doxycycline: Catheter is drained then Doxycycline 500 mg placed in the catheter. Catheter is capped for 1 hour and then drained again.
  Phone Calls: After th
Arm/Group | Indwelling Pleural Catheters (Randomized to Saline) | Indwelling Pleural Catheters Plus Doxycycline (Randomized to R
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Due to slow accrual and the design of the study the protocol was terminated and Adverse Events was not collected.
Arm/Group | Indwelling Pleural Catheters (Randomized to Saline) | Indwelling Pleural Catheters Plus Doxycycline (Randomized to R
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to slow accrual and the design of the study the protocol was terminated and no analysis or adverse event was reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT02623959/Prot_SAP_000.pdf